CLINICAL TRIAL: NCT04776473
Title: Open Versus Closed Treatment of Intra-articular Fractures of the Mandibular Condyle: a Multicentre Randomized Controlled Trial
Brief Title: Treatment of Intra-articular Fractures of the Mandibular Condyle
Acronym: FIAC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP180606; 2019-A00252-55 (Other: IDRCB)
Record Dates: First submitted 2021-02-17; First posted 2021-03-01 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Intra-articular Fracture of the Mandibular Condyle
Keywords: intra-articular fracture; mandibular condyle; surgical treatment; conservative treatment
MeSH Terms: conditions — Intra-Articular Fractures | interventions — Open Abdomen Techniques; Surgical Procedures, Operative; Conservative Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open (i.e. surgical) treatment (Experimental): This includes reduction and internal fixation of the fracture (ORIF) performed using the preferred surgical approach and bone implants of the including centre that could be associated with one or several items among the following:
  * physical therapy based on exercises done by the patient himself
  * physical therapy performed by a specialized/non-specialized physical therapist
  * arch bars / screws / splint use for transient MMF
  * arch bars / screws / splint use for passive mobilization of the mandible
  Interventions: Procedure: Open treatment
- Closed (i.e. conservative) treatment (Other): To date, there is no consensus on which procedures should be used in case of conservative treatment, which may vary between centres and, for a same centre, between patients. This includes one or several items among the following:
  * physical therapy based on exercises done by the patient himself
  * physical therapy performed by a specialized/non-specialized physical therapist
  * arch bars / screws / splint use for transient maxillo-mandibular fixation (MMF) (15 days max)
  * arch bars / screws / splint use for passive mobilization of the mandible
  Interventions: Other: Closed treatment

INTERVENTIONS:
Procedure: Open treatment — Open (i.e. surgical) treatment will be performed following the usual practice of the including centre adopting a pragmatic approach.
  Other Names: Surgical treatment
  Arms: Open (i.e. surgical) treatment
Other: Closed treatment — Closed (i.e. conservative) treatment will be performed following the usual practice of the including centre adopting a pragmatic approach.
  Other Names: Conservative treatment
  Arms: Closed (i.e. conservative) treatment

SUMMARY:
Intra-articular fractures of the mandibular condyle ((IAFC) are usually treated by means of physical therapy with or without transient maxillo-mandibular fixation (conservative or closed treatment). However, this can lead to incomplete manducatory function recovery due to limited mandibular mobility. During the last 15 years, a growing interest has emerged for open (surgical) treatment of these fractures. Although there is more and more evidence suggesting that the open treatment may be the treatment of choice for selected cases of subcondylar fractures, the best option remains controversial for high condylar fractures.

The primary objective of the trial is to compare mandibular mobility at 3 months post-treatment between open (surgical) and closed (conservative) treatment of intra-articular fracture (high fracture) of the mandibular condyle.

This study is an open multicenter randomized controlled trial with 2 parallel arms. Eligible patients will be randomized 1 :1 between open and closed-treatment group.

DETAILED DESCRIPTION:
The mandibular condyle is one of the most frequent locations of facial fractures. It can lead to severe functional impairment if the occlusion is not properly restored and the mandibular mobility not recovered totally or within an acceptable range. Most frequent sequels of these fractures include limitation of mandibular movements resulting in limited mouth opening, occlusal disturbance causing chewing malfunction, chronic pain, chronic temporo-mandibular joint (TMJ) disorder and facial asymmetry. The risk of permanent limited mouth opening is even higher when the fracture is located inside the TMJ. Although the superiority of surgical treatment is now widely accepted for low-level fractures of the condylar unit (i.e., extra-articular fractures) the treatment of fractures involving the TMJ in adult patients is still controversial.

Treatment principles in these fractures can be ranked in two groups: closed and open treatments. Closed treatment - also called closed reduction or conservative treatment - consists in prolonged physical therapy frequently associated with transient maxillo-mandibular fixation (MMF). Open treatment consists in open reduction and internal fixation of the fracture (ORIF).

No randomized controlled trial has ever evaluated the superiority of open versus closed treatment, and treatment strategy for IAFC remains a matter of ongoing debate.

The primary objective of this trial is to compare mandibular mobility at 3 months post-treatment between open (surgical) and closed (conservative) treatment of intra-articular fracture (high fracture) of the mandibular condyle.

The secondary objectives are to compare between open (surgical) and closed (conservative) treatments:

At 3 weeks, 6 weeks, 3 months, 6 months, and 12 months post-treatment:

* maximal mouth opening (in mm)
* maximal mandibular protrusion (in mm),
* maximal lateral excursion (in mm),
* lateral deviation of the mandible during mouth opening
* occlusal disturbance evaluated by both the patient and the surgeon
* pain using a visual analog scale
* subjective functional impairment as assessed by the Mandibular Function Impairment Questionnaire

Overall:

* duration of sick leave
* time to normal activity recovery (social activities, eating, sports) We will also evaluate compliance with the intervention. This trial is an open multicenter randomized controlled trial with 2 parallel arms. Eligible patients will be randomized 1 :1 between open and closed-treatment group.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≥18 y-o) < 85 years
2. Displaced non-comminuted intra-articular fracture of the mandibular condyle (IAFC) as defined by a fracture line above a horizontal line tangent to the mandibular notch
3. Objectifiable induced malocclusion and/or ramus shortening ≥2 mm on CT-scan (a ramus shortening ≥2 mm on CT-scan is necessary in case of other associated mandibular or occluso-facial fractures)
4. Unilateral or bilateral fracture
5. Isolated or associated with other facial / extra-facial skeleton / dental / soft tissue lesions
6. Treatment within 14 days post trauma
7. Affiliation to a social security regime (excepted AME)
8. Written informed consent

Exclusion Criteria:

1. Contraindication to surgical treatment (for any medical or anatomical reason, like comminuted fracture for instance)
2. Major teeth loss or edentulous patient (occlusion impossible to assess)
3. History of mandibular fracture
4. History of temporo-mandibular joint (TMJ) disorder
5. Dentofacial dysmorphosis causing significant malocclusion
6. Predictable inability to comply with the follow-up
7. Unconsciousness / severe polytrauma
8. Participation in another interventional study

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-05-03 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Maximal mouth opening (in mm) at 3 months | 3 months (+/-10 days)
  It will be obtained by measuring the interincisal distance at maximum mouth opening with a caliper or a ruler. The patient will be first asked to open the mouth as widely as possible for 3 seconds and to rest for 5 seconds. This sequence will be repeated 2 times and at the third repetition the patient will keep his/her mouth opened while the physician will measure inter-incisal distance

SECONDARY OUTCOMES:
Maximal mouth opening (in mm) | 3 weeks (+/- 7 days), 6 weeks (+/-7 days), 6 months (+/-20 days) and, 12 months (+/- 30 days) post-treatment
  Measured following the method described for primary outcome.
Maximal mandibular protrusion (in mm) | 3 weeks (+/- 7 days), 6 weeks (+/-7 days), 3 months (+/-10 days), 6 months (+/-20 days) and, 12 months (+/- 30 days) post-treatment
  - Maximal mandibular protrusion in mm measured with a caliper or with a ruler, asking the patient to move the mandible as far as possible in the forward direction while keeping a slight contact between the dental arches. This measure will be done only after repetition of mouth opening and measurement of the maximum mouth opening, which will warm up mandibular mobilization
Maximal lateral excursion (in mm) | 3 weeks (+/- 7 days), 6 weeks (+/-7 days), 3 months (+/-10 days), 6 months (+/-20 days) and, 12 months (+/- 30 days) post-treatment
  Maximal lateral excursion in mm measured with a caliper or with a ruler, asking the patient to move the mandible as far as possible in the right and left directions while keeping a slight contact between the dental arches. These measurements will be done only after repetition of mouth opening and measurement of the maximum mouth opening, which will warm up mandibular mobilization
Lateral deviation of the mandible during mouth opening | 3 weeks (+/- 7 days), 6 weeks (+/-7 days), 3 months (+/-10 days), 6 months (+/-20 days) and, 12 months (+/- 30 days) post-treatment
  Lateral deviation of the mandible during mouth opening will be ranked as straight, right, or left. This observation can be made during the first measurement of mandibular opening
Occlusal disturbance reported by the patient | 3 weeks (+/- 7 days), 6 weeks (+/-7 days), 3 months (+/-10 days), 6 months (+/-20 days) and, 12 months (+/- 30 days) post-treatment
  The patient will be asked to describe how his/her teeth touch as referring to his/her previous occlusion. He/she will rank his/her occlusion as:
  * not modified
  * slightly modified as compared to before the trauma but with no significant disturbance
  * significantly disturbed
Occlusal disturbance evaluated by the surgeon | 3 weeks (+/- 7 days), 6 weeks (+/-7 days), 3 months (+/-10 days), 6 months (+/-20 days) and, 12 months (+/- 30 days) post-treatment
  The surgeon will ask the patient to bite and describe the occlusion as:
  * Not modified
  * Open bite: barely detectable (right / anterior / left) or clearly detectable (right / anterior / left)
  * Premature contact: barely detectable (right / anterior / left) or clearly detectable (right / anterior / left)
Evaluation of pain using a visual analog scale | 3 weeks (+/- 7 days), 6 weeks (+/-7 days), 3 months (+/-10 days), 6 months (+/-20 days) and, 12 months (+/- 30 days) post-treatment
  The patient will be asked to rate his/her maximum pain in the last 2 days on a visual analog scale, 0 representing no pain and 10 representing the worst pain imaginable.
  For bilateral fractures, the pain will be assessed separately on each side.
Subjective functional impairment evaluated by the patient using the Mandibular Function Impairment Questionnaire (MFIQ) | 3 weeks (+/- 7 days), 6 weeks (+/-7 days), 3 months (+/-10 days), 6 months (+/-20 days) and, 12 months (+/- 30 days) post-treatment
  The Mandibular Function Impairment Questionnaire (MFIQ) consisting in 17 items, rated between 0 and 4, which describes the difficulty in several common movement/activities involving the mandible (see questionnaire 1).
Duration of sick leave | From treatment until 12 months
Time to normal activity recovery | Every week from week 1 to 6, every 2 weeks from week 8 to 12, and every month from month 4 to 12
  Patient will asked on return to work and to normal daily activities (social activities, eating, sports)
Compliance with the intervention - Number of appointments with a physical therapist | Every week from week 1 to 6, every 2 weeks from week 8 to 12, and every month from month 4 to 12
  The patient will fill in a notebook the number of appointments with a physical therapist since last patient report.
Compliance with the intervention - Number of self-training sessions | Every week from week 1 to 6, every 2 weeks from week 8 to 12, and every month from month 4 to 12
  The patient will fill in a notebook the number of the number of self-training sessions since last patient report
Compliance with the intervention - Duration of permanent MMF | Every week from week 1 to 6, every 2 weeks from week 8 to 12, and every month from month 4 to 12
  The patient will fill in a notebook the number of permanent MMF since last patient report
Compliance with the intervention - Duration of transient MMF | Every week from week 1 to 6, every 2 weeks from week 8 to 12, and every month from month 4 to 12
  The duration of permanent MMF the duration of transient MMF since last patient report
Compliance with the intervention - Duration of application of mobilization elastic band | Every week from week 1 to 6, every 2 weeks from week 8 to 12, and every month from month 4 to 12
  The patient will fill in a notebook the duration of application of mobilization elastic band.
Compliance with the intervention - Average and Maximal pain | Every week from week 1 to 6, every 2 weeks from week 8 to 12, and every month from month 4 to 12
  The patient will fill in a notebook the average and maximal pain rate since last patient report

CONTACTS AND LOCATIONS:
Overall Officials: Thomas SCHOUMAN, MD, Principal Investigator — AP-HP - Hôpital Pitié-Salpêtrière
Locations (7):
- France (7):
  - CHU Angers, Angers
  - Hôpital Annecy Genevois, Annecy
  - APHM - Hôpital de la Conception, Marseille
  - CHU de Nantes, Nantes
  - Hôpital Pitié-Salpêtrière, Paris
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - CHU Purpan - Hôpital Pierre-Paul Riquet, Toulouse

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients. Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal